CLINICAL TRIAL: NCT07303283
Title: Becotatug Vedotin Versus Capecitabine as Adjuvant Therapy for Locoregional Advanced Nasopharyngeal Carcinoma: a Multicentre, Open-label, Parallel-group, Randomised, Controlled, Phase 2 Trial
Brief Title: Becotatug Vedotin as Adjuvant Therapy For High-risk Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kai Hu (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); First People's Hospital of Yulin (Other); Guigang People's Hospital (Other); Hainan Cancer Hospital (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); Affiliated Hospital of Youjiang Medical University for Nationalitie (Unknown); Lingshan people's Hospital (Unknown); People's Hospital of Guangxi Zhuang Autonomous Region (Other); LiuZhou People's Hospital (Other); The Third people's hospital of Hechi (Unknown); the second People's Hospital of qinzhou (Unknown)
Responsible Party: Sponsor-Investigator, Kai Hu, professor, Guangxi Medical University
Organization: Guangxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GuangxiMUHK5
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Nasopharyngeal Carcinoma (NPC); Locoregionally Advanced Nasopharyngeal Carcinoma; Adjuvant Therapy
Keywords: Nasopharyngeal Carcinoma; Adjuvant therapy; Becotatug Vedotin; Capecitabine
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant Becotatug Vedotin (Experimental): Adjuvant therapy with Becotatug Vedotin
  Interventions: Drug: Becotatug Vedotin
- control (Other): Adjuvant therapy with capecitabine
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: Becotatug Vedotin — This group will receive Becotatug Vedotin at a dose of 2.3 mg/kg on day 1 of each 3-week cycle for a total of 3 cycles.
  Arms: Adjuvant Becotatug Vedotin
Drug: capecitabine — Receive capecitabine at 1000 mg/m² twice daily on days 1-14 of each 3-week cycle for 8 cycles.
  Arms: control

SUMMARY:
This is a phase 2, multicentre, open-label, randomised, controlled trial with a parallel-group design. The study aims to compare the efficacy and safety of Becotatug Vedotin and capecitabine as an adjuvant therapy in patients with high-risk locoregionally advanced nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
Eligible patients with high-risk locoregionally advanced nasopharyngeal carcinoma (NPC), staged as T4 N1 M0 or T any N2-3 M0, who have completed curative chemoradiotherapy, will be randomized to either an adjuvant capecitabine group or an adjuvant Becotatug Vedotin group. The experimental group will receive Becotatug Vedotin at a dose of 2.3 mg/kg on day 1 of each 3-week cycle for 3 cycles. The control group will receive capecitabine at 1000 mg/m² twice daily on days 1-14 of each 3-week cycle for 8 cycles. The primary endpoint is failure-free survival (FFS). Secondary endpoints include overall survival (OS), distant metastasis-free survival (D-MFS), locoregional failure-free survival (LR-FFS), and treatment-emergent adverse events. All efficacy analyses will be performed on an intention-to-treat (ITT) basis. Safety analyses will be conducted in the safety population, defined as all patients who received at least one dose of the assigned study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-keratinizing nasopharyngeal carcinoma(WHO II/III).
2. Original clinical staged as TanyN2-3M0 or T4N1M0 (according to AJCC 9th edition), with no evidence of distant metastasis.
3. ECOG performance status ≤1.
4. Induction and concurrent chemoradiotherapy with the recommended regimen have been completed.
5. No later than 6 weeks after the completion of the last radiotherapy treatment.
6. Adequate hematologic (neutrophil count > 1.5×10^9/L, hemoglobin > 90g/L and platelet count > 100×10^9/L), hepatic (alanine aminotransferase, aspartate aminotransferase ≤ 1.5×ULN, bilirubin ≤ 1.5×ULN, alkaline phosphatase < 2.5×ULN) and renal function (creatinine clearance > 50 ml/min)
7. Patients must be informed of the investigational nature of this study and give written informed consent.
8. Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug.

Exclusion Criteria:

1. Patients who could not tolerate or were allergic to Becotatug Vedotin.
2. Patients with severe chronic or active infection that must be treated with systemic antibacterial, antifungal, or antiviral therapy before randomization, including but not limited to tuberculosis infection.
3. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
4. Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
5. Interstitial lung disease or pneumonia requiring oral or intravenous steroid therapy within 1 year.
6. Patients who are known to be intolerant or sensitive to any therapeutic agents.
7. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
failure-free survival | 2 years
  calculated from the date of randomisation to the date of locoregional failure, distant failure, or death from any cause, whichever occurred first

SECONDARY OUTCOMES:
overall survival | 2 years
  calculated from the date of randomisation to death
distant metastasis-free survival | 2 years
  calculated from the date of randomisation to the first distant metastasis
Locoregional failure-free survival | 2 years
  calculated from the date of randomisation to the first locoregional failure
treatment-related adverse events (AEs) | 5 years
  graded according to NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China